CLINICAL TRIAL: NCT01532804
Title: A Multicenter Randomized Phase 2 Trial to Evaluate the Triplet Combination of Raltitrexed, Oxaliplatin and Bevacizumab Versus FOLFOX6 Plus Bevacizumab in Second-line Treatment of Metastatic Colorectal Cancer
Brief Title: 2nd-line Treatment of Metastatic Colorectal Cancer
Acronym: BEVATOMOX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: too slow recruiting
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEVATOMOX; 2010-023447-15 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Unresectable metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): FOLFOX6 + bevacizumab (D1=D15, 12 cycles)
  Interventions: Drug: bevacizumab, oxaliplatin and 5FU combination
- Arm B (Experimental): Raltitrexed + Oxaliplatin + Bevacizumab (D1=D21, 8 cycles)
  Interventions: Drug: Bevacizumab, oxaliplatin and raltitrexed combination

INTERVENTIONS:
Drug: bevacizumab, oxaliplatin and 5FU combination — Bevacizumab 5 mg/kg administered as an iv infusion for 1h30, then for 1h and for 30 min. at the following cycles, respectively.
  Oxaliplatin 85 mg/m² administered as an iv infusion for 2h Elvorine 200 mg/m² administered as an iv infusion for 2h 5FU 400 mg/m2 bolus then 5FU 2,400 mg/m² iv infusion for 46h D1=D15 (12 cycles)
  Arms: Arm A
Drug: Bevacizumab, oxaliplatin and raltitrexed combination — Bevacizumab 7.5 mg/kg administered as an iv infusion for 1h30, then administered for 1h and 30 min at the following cycles, respectively.
  Oxaliplatin 130 mg/m² administered as an iv infusion for 2h Raltitrexed 3 mg/m² administered as an iv infusion for 15 min
  Arms: Arm B

SUMMARY:
This phase 2 trial aims to evaluate the continued use of bevacizumab with raltitrexed and oxaliplatin combination versus FOLFOX6 plus bevacizumab in patients with metastatic colorectal cancer whose disease has progressed after irinotecan-based chemotherapy.

DETAILED DESCRIPTION:
Eligible patients are randomly allocated to receive either bevacizumab with raltitrexed and oxaliplatin combination or bevacizumab with FOLFOX 6 combination. Random allocation schedule is performed using a minimization technique for the following stratification factors:

* Center
* Number of metastatic sites: 1 versus > 1
* Bevacizumab-based first-line therapy: Yes versus No

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal cancer
* Resected or asymptomatic primary tumor
* Metastatic colorectal cancer not eligible for curative surgery
* No major surgery within four weeks of the start of study treatment
* At least one target lesion unidimensionally measurable on cross-sectional imaging according to RECIST criteria (v1.1)
* Disease progression after failure of irinotecan-based chemotherapy
* Bone metastases are allowed if there is at least one other measurable metastatic site
* CT scan of the abdomen, chest and pelvis within 3 weeks of the start of study treatment
* WHO PS ≤ 2
* Platelet count >= 100,000 mm3
* Hemoglobin > 10g/dl
* Bilirubin < 1.5 ULN, AST/ALT < 5 ULN
* Serum creatinine < 1.5 ULN, creatinine clearance > 60 ml/min (Cockcroft)
* A time period of 4 weeks should be respected between the end of previous treatments and study enrollment
* Negative pregnancy test in women of childbearing potential
* Male or female using an effective contraceptive method
* Absence of known or symptomatic brain metastases
* Life expectancy > 3 months
* Informed consent signed prior any study specific procedures

Exclusion Criteria:

* Prior raltitrexed-based chemotherapy
* Prior oxaliplatin-based chemotherapy (except for adjuvant treatment completed for more than 6 months)
* Uncontrolled arterial hypertension defined as systolic pressure > 150 mm Hg or diastolic pressure > 100 mm Hg
* Malignant hypertension or hypertensive encephalopathy
* Myocardial infarction, pulmonary embolism, or severe vascular disease within 6 months prior to study entry
* Hemorrhagic diathesis or significant pathology of coagulation
* Peripheral neuropathy grade>2 (NCI-CTC v4.0)
* Hemoptysis < 1 month
* Venous access device (PAC) or any other minor surgery such as a biopsy within the last 7 days
* Symptomatic brain metastases or carcinomatous meningitis
* History or presence of other cancer within the past 5 years (except curatively treated nonmelanoma skin cancer and in situ cervical cancer)
* Severe bacterial or fungal infection (Grade > 2 NCI-CTCAE v.4.0)
* Known or suspected sensitivity to one of the study drugs
* Pregnant or breastfeeding women
* Previous enrollment in an investigational drug study within the last 4 weeks
* Psychological, social, geographical disorders or any other condition that would preclude study compliance (treatment administration and study follow-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 6 months
  DFS is estimated from the date of randomization until the first date of objectively documented event or death

SECONDARY OUTCOMES:
Treatment-related toxicity | 6 months
  Treatment-related toxicity is evaluated according to the NCI-CTCAE v.4 criteria.
Objective response rate | Every 9 weeks
  Objective response rate is evaluated according to the RECIST V 1.1 criteria.
Overall survival | unk
  OS is estimated from the date of randomization until the date of death from any cause
Cost-effectiveness study | 6 months
  The cost-effectiveness study includes the number of hospital stays (treatment and toxicity), the global cost of treatments, and the cost of hospital stays due to treatment-induced toxicity
Quality of life by using the quality of life questionnaire score | 6 months
  Quality of life is measured using the QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Samalin-Scalzi, MD, Principal Investigator — Val d'Aurelle Cancer Institute
Locations (1):
- Val d'Aurelle Cancer Institute, Montpellier, France

REFERENCES:
- [Derived] Samalin E, Senellart H, Thezenas S, Jacquot S, Ellis S, Akouz FK, Fiess C, Ramdani M, Portales F, Assenat E, Ychou M, Mineur L, Mazard T. The BEVATOMOX phase II trial: raltitrexed/oxaliplatin/bevacizumab vs mFOLFOX6/bevacizumab in 2nd-line metastatic colorectal cancer. Oncologist. 2026 Jan 14:oyag006. doi: 10.1093/oncolo/oyag006. Online ahead of print. PMID 41537257